CLINICAL TRIAL: NCT00103740
Title: Randomized, Double-Blind, Safety and Efficacy Trial With Intravenous Zoledronic Acid for the Treatment of Paget's Disease of Bone Using Risedronate as a Comparator, Including an Extended Observation Period
Brief Title: Safety and Efficacy Trial With Zoledronic Acid for the Treatment of Paget's Disease of Bone, Including an Extended Observation Period
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446H2305; ZOL446K2305 (Other: Novartis Pharmaceuticals); NCT00051649 (obsolete NCT alias)
Record Dates: First submitted 2005-02-14; First posted 2005-02-15 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Paget's Disease of Bone
Keywords: Zoledronic acid, risedronate, Paget's disease of bone
MeSH Terms: conditions — Osteitis Deformans | interventions — Zoledronic Acid; Risedronic Acid; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Zoledronic acid and placebo to risedronate (Experimental): Participants received zoledronic acid 5.0 mg i.v. infusion one dose, 60 days of oral placebo to risedronate, calcium 500mg bid and vitamin D 400 to 1000 IU daily during the core period, and received only calcium and vitamin D supplements during the extended observation period.
  Interventions: Drug: zoledronic acid; Drug: Placebo to risedronate; Drug: Calcium and vitamin D supplements
- Risedronate and placebo to zoledronic acid (Active Comparator): Participants received 60 days of oral risedronate 30 mg, one i.v. infusion of placebo to zoledronic acid infusion, calcium 500mg bid and vitamin d 400 to 1000 IU daily during the core period, and received only calcium and vitamin D supplements during the extended observation period.
  Interventions: Drug: placebo to zoledronic acid; Drug: Risedronate; Drug: Calcium and vitamin D supplements

INTERVENTIONS:
Drug: zoledronic acid — 5 mg zoledronic acid in 5 mL of sterile water for infusion
  Arms: Zoledronic acid and placebo to risedronate
Drug: placebo to zoledronic acid — 5 mL of sterile water for infusion
  Arms: Risedronate and placebo to zoledronic acid
Drug: Risedronate — 30mg oral tablets overencapsulated to match the placebo capsules
  Arms: Risedronate and placebo to zoledronic acid
Drug: Placebo to risedronate — oral capsules
  Arms: Zoledronic acid and placebo to risedronate
Drug: Calcium and vitamin D supplements — Calcium and vitamin D supplements were supplied

SUMMARY:
The primary objective of this core study was to show non-inferiority of zoledronic acid to risedronate, with respect to the proportion of patients who achieved therapeutic response. The extended observation period included participants of the core study who responded to treatment.

ELIGIBILITY:
Inclusion Criteria:

* 30 years or older
* SAP 2 times ULN
* Confirmed diagnosis of Paget's disease of the bone (by x-ray, magnetic resonance imaging, computerized tomography, radioisotope imaging, etc.).
* 90 days washout calcitonin
* 180 day washout bisphosphonate

Exclusion Criteria:

* Allergic reaction to bisphosphonates
* History of upper GI disorders
* History of iritis, uveitis
* Calculated creatinine clearance < 30 ml/min at baseline
* Evidence of vitamin D deficiency

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2002-04; Primary Completion 2003-12 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (41):
- United States (10):
  - Novartis Investigative site, Tucson, Arizona
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Syracuse, New York
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Madison, Wisconsin
- Australia (5):
  - Novartis Investigative Site, Fitzroy
  - Novartis Investigative Site, Kogarah
  - Novartis Investigative site, Newcastle
  - Novartis Investigative Site, Parkville
  - Novartis Investigative site, St Leonards
- Belgium (2):
  - Novartis Investigative site, Brussels
  - Novartis Investigative Site, Ghent
- Novartis Investigative Site, Montreal, Canada
- France (7):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Dreux
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Wirzburg
- Novartis Investigative site, Christchurch, New Zealand
- Novartis Investigative site, Cape Town, South Africa
- Spain (6):
  - Novartis Investigative site, Barcelona
  - Novartis Investigative site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative site, Santiago de Compostela
  - Novartis Investigative Site, Valencia
- United Kingdom (3):
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative site, Oxford

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 371 patients were screened. 185 patients were randomized.
Period: Period 1 - Core
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Started | 92 | 93
Completed | 85 | 89
Not Completed | 7 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 3 | 2
Not completed — Patient withdrew consent | 3 | 2
Period: Period 2 - Extended Observation Period
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Started | 78 | 63
Completed | 9 (Includes patients retreated for Paget's disease and patients discontinued when sponsor ended study) | 27 (Includes patients retreated for Paget's disease and patients discontinued when sponsor ended study)
Not Completed | 69 | 36
Not completed — Lost to Follow-up | 7 | 6
Not completed — Withdrew for nonclinical reason | 21 | 13
Not completed — Clinical reason other than Paget's | 5 | 6
Not completed — Death | 6 | 2
Not completed — Amendment 6 informed consent not signed | 30 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid | Total
Number analyzed (Participants) | 92 | 93 | 185
Age Continuous [Mean (Standard Deviation); unit: years] | 71.3 (9.42) | 68.2 (11.15) | 69.8 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 36 | 66
  Male | 62 | 57 | 119

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Had Therapeutic Response at 6 Months
Description: A therapeutic response was defined as a reduction of at least 75% from baseline (Visit 1) in serum alkaline phosphatase (SAP) excess (difference between measured level and midpoint to the normal range) or normalization of SAP at the end of six months.
Time Frame: Baseline, 6 months
Population: Modified intent to treat population: all randomized patients with both baseline and at least one post-baseline serum alkaline phosphatase measurement. Missing values at 6 months were imputed using the last post-baseline measurement prior to 6 months.
Measure: Number; unit: participants
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 88 | 89
participants | 84 | 67

2. Secondary Outcome: Relative Change in Serum Alkaline Phosphatase in U/L at Day 28
Description: The percent change in serum alkaline phosphatase from baseline to Day 28 was measured.
Time Frame: Baseline and 28 days
Population: Intent-to-treat population: all randomized patients. Participants with observations at baseline and 28 days were included in this analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 79 | 85
percent change | -49.1 (14.55) | -24.3 (18.19)

3. Secondary Outcome: Relative Change in Serum C-telopeptide (CTx) in ng/mL at Day 10
Description: The percent change in serum C-telopeptide from baseline to Day 10 was measured.
Time Frame: Baseline and day 10
Population: Intent-to-treat population: all randomized patients. Participants with observations at baseline and day 10 were included in this analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 60 | 70
percent change | -74.2 (123.73) | -40.1 (34.70)

4. Secondary Outcome: Relative Change in Urine α-CTx in ug/mmol at Day 10
Description: The percent change in urine α-CTx from baseline to Day 10 was measured.
Time Frame: Baseline and day 10
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 67 | 70
percent change | -87.5 (39.33) | -28.7 (68.22)

5. Secondary Outcome: Time to First Therapeutic Response
Description: Therapeutic response was defined as a reduction of at least 75% from baseline in serum alkaline phosphatase excess (difference between measured level and midpoint to the normal range) or normalization of serum alkaline phosphatase.
Time Frame: 182 days
Population: Intent-to-treat population: all randomized patients.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 92 | 93
days | 64 [33 to 65] | 91 [64 to 181]

6. Secondary Outcome: Number of Patients Who Achieved Serum Alkaline Phosphatase Normalization at Day 28
Description: Normalization of serum alkaline phosphatase occurred if the serum alkaline phosphatase measurement fell within the normal range. Central laboratory reference ranges for serum alkaline phosphatase: 31-110 U/L (female & male 20-58 years) and 35-115 U/L (female & male >58 years).
Time Frame: Day 28
Population: Intent-to-treat population: all randomized patients. Participants with observations at day 28 were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 88 | 88
participants | 8 | 1

7. Secondary Outcome: Change in Pain Severity at Day 182
Description: Change in pain severity score from Brief Pain Inventory-Short Form (BPI-SF). This scale values are 0 to 10, a lower score means little to no pain while a higher score means greater pain.
Time Frame: Baseline and day 182
Population: Intent-to-treat population: all randomized patients. Participants with observations at baseline and day 182 were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 50 | 46
units on a scale | -0.5 (1.74) | -0.1 (2.02)

8. Secondary Outcome: Change in Pain Interference at Day 182
Description: Change in pain interference score from Brief Pain Inventory-Short Form (BPI-SF). This scale values are 0 to 10, a lower score means little to no pain while a higher score means greater pain.
Time Frame: Baseline and day 182
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 49 | 45
units on a scale | -0.5 (1.97) | 0.0 (1.89)

9. Secondary Outcome: Number of Participants With a Loss of Therapeutic Response During the Extended Observation Period
Description: Extended observation period. A therapeutic response is defined as a reduction of at least 75% from baseline in serum alkaline phosphatase excess or normalization of serum alkaline phosphatase.
Time Frame: 8 years was the maximum
Population: Extended modified Intent-to-treat population: patients who had at least one serum alkaline phosphatase measurement during the extension period.
Measure: Number; unit: participants
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 78 | 63
participants | 10 [2218 to NA] | 42 [344 to 1605]

10. Secondary Outcome: Number of Participants With a Partial Disease Relapse During the Extended Observation Period
Description: Extended observation period. A partial disease relapse was defined as an increase in serum alkaline phosphatase >= 50% from the serum alkaline phosphatase measurement at Month 6 and at least 1.25 times the upper normal limit.
Time Frame: 8 years was the maximum
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 78 | 63
participants | 9 [2218 to NA] | 37 [373 to 1652]

11. Secondary Outcome: Number of Participants With a Disease Relapse During the Extended Observation Period
Description: Extended observation period. A disease relapse was defined as the occurrence of a serum alkaline phosphatase level that was >= 80% of baseline serum alkaline phosphatase value.
Time Frame: 8 years was maximum
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 78 | 63
participants | 0 [NA to NA] | 15 [1084 to NA]

ADVERSE EVENTS:
Description: The safety population consisted of all randomized patients who were exposed to study drug.
Groups:
- Zoledronic Acid: Participants received zoledronic acid 5.0 mg i.v. infusion one dose, 60 days of oral placebo to risedronate, calcium 500mg bid and vitamin D 400 to 1000 IU daily during the core period, and received only calcium and vitamin D supplements during the extended observation period.
- Risedronate: Participants received 60 days of oral risedronate 30 mg, one i.v. infusion of placebo to zoledronic acid infusion, calcium 500mg bid and vitamin d 400 to 1000 IU daily during the core period, and received only calcium and vitamin D supplements during the extended observation period.
Arm/Group | Zoledronic Acid | Risedronate
Serious Adverse Events (participants affected / at risk) | 4/88 | 3/90
Other Adverse Events (participants affected / at risk) | 40/88 | 28/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=88) | Risedronate (N=90)
Chest pain (General disorders) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=88) | Risedronate (N=90)
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 6 | 3
Fatigue (General disorders) | 6 | 2
Influenza like illness (General disorders) | 13 | 6
Influenza (Infections and infestations) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Dizziness (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.